CLINICAL TRIAL: NCT06703580
Title: Intrathecal Hyperbaric Prilocaine in Adult Patients Undergoing Knee Arthroscopy, a Randomized Controlled Trail
Brief Title: Using Three Different Doses of Hyperbaric Prilocaine 2% Local Anaesthetic ( 40,50 and 60mg ),Through Spinal Anaesthesia in Knee Arthroscopy Patients to Compare Time to Void
Acronym: Prilocaine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa mahmoud bahaa eldin mohamed taha, lecturer of anaesthesia , surgical ICU and pain -cairo university, Cairo University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Health Services Research
Other Study IDs: MS-213-2023
Record Dates: First submitted 2024-11-05; First posted 2024-11-25 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Time to First Void After Spinal Anaesthesia
Keywords: prilocaine; intrathecal; day case; arthroscopy; time to void

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- arm 40 (Active Comparator)
  Interventions: Drug: Hyperbaric prilocaine 2% 40 mg
- arm 50 (Active Comparator): this arm will include 50 patients who will receive intrathecal hyperbaric prilocaine 2% in the dose of 50 mg.
  Interventions: Drug: hyperbaric prilocaine 2% 50 mg
- arm 60 (Active Comparator): this arm will include 50 patients who will receive intrathecal hyperbaric prilocaine 2% in the dose of 60 mg
  Interventions: Drug: hyperbaric prilocaine 2% 60 mg

INTERVENTIONS:
Drug: Hyperbaric prilocaine 2% 40 mg — this arm will include 50 patients who will receive intrathecal hyperbaric prilocaine 2% in a dose of 40 mg.
  Arms: arm 40
Drug: hyperbaric prilocaine 2% 50 mg — comparison of 3 different doses of prilocaine
  Arms: arm 50
Drug: hyperbaric prilocaine 2% 60 mg — this study compare 3 different doses of prilocaine
  Arms: arm 60

SUMMARY:
The goal of this randomised trial is to use a short acting local anaesthetic drug (hyperbaric prilocaine 2%) which is beneficial in short operations which are performed as a day case surgery.

in this study the investigators will use 3 different doses of prilocaine 2% (40,50 or 60 mg ) intrathecal (in spinal anaesthesia) in participants undergoing arthroscopy on the knee.

the primary outcome is to compare time to micturate (go to the bathroom) between the three groups .

the secondary outcomes are:

* time to recovery of the motor and sensory block
* time to discharge from post anesthesia care unit
* any complications ; itching, lowered blood pressure, nausea and vomiting.

ELIGIBILITY:
Inclusion Criteria:

All patients (male/female, American Society of Anesthesiologists physical status I-II, age: 18-60 years) undergoing knee arthroscopy will be eligible for the study. -

Exclusion Criteria:

1. Coagulopathy and other bleeding disorders (INR more than 1.4 and platelet less than 80000)
2. Patient refusal.
3. Infection at the site of injection.
4. Allergies against prilocaine.
5. Increased intracranial pressure.
6. Severe MS and AS.
7. Sever hypovolemia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-12-27 (Actual); Study Completion 2026-02-08 (Actual)

PRIMARY OUTCOMES:
Time to void; time from spinal anaesthesia to first void | from time of spinal anaesthesia as a start point till time for the participant to get up and micturate on his own (time to first void) assessed up to 4 hours postoperative
  we will measure the time from spinal anaesthesia to first void and compare that in the 3 groups with different doses of hyperbaric prilocaine 2% (40,50 and 60 mg) to see which group has the least time to void and so early ambulation in a day case surgery of knee arthroscopy.

SECONDARY OUTCOMES:
Motor block regression time | The motor block will be assessed 10 min after intrathecal injection as a start point and every 30 minutes until recovery of full motor power (bromage 0) up to 4 hours postoperative
  Motor block will be measured by using modified bromage score, 0 = no motor block; 1 = unable to lift the extended leg in the hips; 2 = unable to flex hips and knees but still able to flex ankles; 3 = complete motor block of the lower extremity.
sensory regression time | sensory regression time will be measured 10 minutes after intrathecal block (as a start point) and then every 30 minutes until regression to two dermatomes intra-operative and until 4 hours post-operative.
  sensory regression time will be assessed thermally with an ice- filled plastic tube and by using wooden toothpick.
heart rate | heart rate will be measured in the form of beats /min from the start of operation and every 5 minutes till the end of operation
mean arterial pressure | mean arterial pressure (MAP) will be measured in mmhg every 5 minutes from the start of operation till the end of operation
Incidence of complications | incidence of complications will be recorded from the start of operation till discharge from post anaesthesia care unit (PACU) assessed up to 4 hours
  incidence of hypotension, bradycardia, nausea, vomiting , headache or pruritis if it occurred or not ( as a yes or no)
Time to discharge from post operative anaesthesia unit (PACU) | time will be recorded from the start of operation till discharge of the participant from PACU after reaching Aldrete score of 10 (up to 4 hours postoperative)

CONTACTS AND LOCATIONS:
Overall Officials: osama M Asad, professor of anaesthesia, Study Chair — Cairo University
Locations (1):
- Kasr Al Ainy Hospital , Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol